CLINICAL TRIAL: NCT04893811
Title: A PHASE 4, OPEN-LABEL, SINGLE-ARM TRIAL TO DESCRIBE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF TRUMENBA(REGISTERED) WHEN ADMINISTERED TO IMMUNOCOMPROMISED PARTICIPANTS ≥10 YEARS OF AGE
Brief Title: Trial to Describe the Safety, Tolerability, and Immunogenicity of Trumenba When Administered to Immunocompromised Participants ≥10 Years of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B1971060; 2018-002588-24 (EudraCT Number)
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Meningococcal Vaccine
Keywords: Meningococcal Vaccine; Meningitis Vaccine; Asplenia; Sickle cell anemia; Complement deficiencies
MeSH Terms: conditions — Anemia, Sickle Cell; Hereditary Complement Deficiency Diseases | interventions — MenB-FHbp vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Bivalent recombinant lipoprotein 2086 vaccine
  Interventions: Biological: Trumenba

INTERVENTIONS:
Biological: Trumenba — Bivalent recombinant lipoprotein 2086 vaccine

SUMMARY:
The aim of this study is to evaluate the safety, tolerability, and immunogenicity of 2 doses of Trumenba® (on a 0- and 6-month schedule) in immunocompromised participants by functionally assessing antibody production in asplenic and complement-deficient individuals ≥10 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥10 years of age at the time of consent.
* Participants with an increased risk for meningococcal disease due to anatomic asplenia or functional asplenia (eg, sickle cell anemia) or complement deficiencies.
* Negative urine pregnancy test for all female participants.

Exclusion Criteria:

* Previous vaccination with any meningococcal serogroup B vaccine.
* Participants who are receiving any allergen immunotherapy with a nonlicensed product or receiving allergen immunotherapy with a licensed product and are not on stable maintenance doses.
* History of microbiologically proven disease caused by N meningitidis or Neisseria gonorrhoeae.
* Significant neurological disorder or history of seizure (excluding simple febrile seizure).
* Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.
* Any confirmed or suspected human immunodeficiency virus infection.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Receipt of immunoglobulin infusion or injection during the 42 days preceding enrollment.
* Current chronic use of systemic antibiotics.
* Previous receipt or current use of complement inhibitors (eg, eculizumab, ravulizumab).
* Participation in other studies involving investigational drug(s) within 28 days prior to study entry and/or during study participation.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Czechia (2):
  - Fakultni Nemocnice Brno - Detska Nemocnice - Klinika Detskych Infekcnich Nemoci Center 3, Brno
  - Fakultni nemocnice v Motole, Prague
- Poland (4):
  - IN-VIVO Sp. z o.o., Bydgoszcz
  - Centrum Badań Klinicznych Jagiellońskie Centrum Innowacji sp. z o.o., Krakow
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Szpital Bielański im. Ks. Jerzego Popiełuszki SPZOZ, Warsaw
- Turkey (Türkiye) (5):
  - Baskent Universitesi Dr. Turgut Noyan Adana Uygulama ve Arastirma Merkezi, Adana, Yüreği̇r
  - Baskent Universitesi Dr. Turgut Noyan Adana Uygulama ve Arastirma Merkezi, Adana
  - Acibadem Adana Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1971060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 53 immunocompromised participants greater than or equal to (>=) 10 years of age with asplenia (anatomic or functional) or complement deficiency were enrolled and received Trumenba on a 2-dose, 0- and 6-month schedule in the Study B1971060 [NCT04893811].
Pre-assignment Details: Historical data from age- and sex-matched healthy participants (randomly selected) from previously completed Phase 3 Study B1971057 (Stage 1) [NCT03135834] was used as a reference for safety and immunogenicity analysis of Trumenba administered in the current Study B1971060 [NCT04893811]. Participants whose historical data was used for reference/control, were not included in enrolment number of the current study.
Groups:
- Trumenba (B1971060): Eligible participants were enrolled and received Trumenba 0.5 milliliter (mL), intramuscularly (IM) on Day 1 of Visit 1 (Month 0, Vaccination 1) and Visit 3 (Month 6, Vaccination 2) in the study B1971060. Vaccination phase was from the date of the first vaccination (Visit 1) through 1 month after the second vaccination (Visit 4) and Follow-up phase was defined as the time from 1 month after the second vaccination (Visit 4) through 6 months after the second vaccination (Visit 5).
- Trumenba (B1971057, Historical Age- and Sex-Matched Control): Age- and sex-matched healthy participants from group 2 or 4 (Trumenba groups) from study B1971057 Stage 1 [NCT03135834] were randomly selected and included in this group. Participants included in this arm were not enrolled in the study, only their historical data was used as a reference. This arm served as a control arm for the study.
Period: Vaccination Phase
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Started | 53 | 51
Vaccination 1 | 53 | 51
Vaccination 2 | 47 | 47
Completed | 47 | 47
Not Completed | 6 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 0 | 1
Not completed — No longer met eligibility criteria | 0 | 1
Period: Follow-up Phase
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Started | 47 | 47
Follow-up Safety Set (B1971060: Follow-up safety set included all participants who received at least 1 dose of study intervention and for whom safety information was available from after Visit 4 up to and including Visit 5. B1971057: Historical data of the age- and sex-matched healthy participants (selected randomly) as reference for current study.) | 44 | 48
Completed | 47 | 46
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: For B1971060: all enrolled participants who received at least 1 dose of the study Intervention. For B1971057: Historical data of the age- and sex-matched healthy participants (selected randomly) as reference for current study.
Groups:
- Trumenba (B1971060): Eligible participants were enrolled and received Trumenba 0.5 mL, IM on Day 1 of Visit 1 (Month 0, Vaccination 1) and Visit 3 (Month 6, Vaccination 2) in the study B1971060. Vaccination phase was from the date of the first vaccination (Visit 1) through 1 month after the second vaccination (Visit 4) and Follow-up phase was defined as the time from 1 month after the second vaccination (Visit 4) through 6 months after the second vaccination (Visit 5).
- Total: Total of all reporting groups
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control) | Total
Number analyzed (Participants) | 53 | 51 | 104
Age, Customized [Count of Participants; unit: Participants]
  2-11 years | 2 | 2 | 4
  12-17 years | 8 | 6 | 14
  18-64 years | 40 | 43 | 83
  65-84 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 30 | 30 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 7 | 7
  Not Hispanic or Latino | 53 | 44 | 97
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 53 | 46 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titer => Lower Limit of Quantitation (LLOQ) for Each of the 4 Primary Neisseria Meningitidis Serogroup B (MnB) Test Strains at Baseline
Description: Four primary MnB strains were PMB80 (A22), PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44). The percentage of participants who achieved an hSBA titer PMB80 (A22) more than or equal to (=>)1:16, and hSBA titer PMB2001 (A56), PMB2001 (B24), and PMB2707 (B44) =>1:8 are reported. Evaluable immunogenicity population (EIP) included all participants who were eligible through 1 month after Vaccination 2, received the study vaccination at Visit 1 and Visit 3 as planned, had blood drawn for assay testing within the required time frames at Visit 1 (before Vaccination 1) and 1 month after Vaccination 2 (28-42 days after Visit 3), had at least 1 valid and determinate assay result 1 month after Vaccination 2, received no prohibited vaccines or medications through Visit 4, and had no major protocol deviations through Visit 4.
Time Frame: Baseline (Before Vaccination 1 on Day 1/Month 0)
Population: B1971060: EIP was analyzed. B1971057: Historical data of the age- and sex-matched healthy participants (selected randomly) as reference for current study, relevant for this outcome measure. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 43 | 44
Percentage of participants
  PMB80 (A22): number analyzed (Participants) | 43 | 42
  PMB80 (A22) | 32.6 [19.1 to 48.5] | 31.0 [17.6 to 47.1]
  PMB2001 (A56): number analyzed (Participants) | 43 | 43
  PMB2001 (A56) | 25.6 [13.5 to 41.2] | 23.3 [11.8 to 38.6]
  PMB2948 (B24): number analyzed (Participants) | 42 | 43
  PMB2948 (B24) | 2.4 [0.1 to 12.6] | 23.3 [11.8 to 38.6]
  PMB2707 (B44) | 9.3 [2.6 to 22.1] | 11.4 [3.8 to 24.6]

2. Primary Outcome: Percentage of Participants With hSBA Titer => LLOQ for Each of the 4 Primary MnB Test Strains at 1 Month After Vaccination 2
Description: Four primary MnB strains were PMB80 (A22), PMB2001 (A56), PMB2948 (B24) and PMB2707 (B44). The percentage of participants who achieved an hSBA titer PMB80 (A22) =>1:16, and hSBA titer PMB2001 (A56), PMB2001 (B24), and PMB2707 (B44) =>1:8 were reported.
Time Frame: 1 Month after Vaccination 2 (Vaccination 2 at Month 6)
Population: B1971060: EIP was analyzed. B1971057: Historical data of the age- and sex-matched healthy participants (selected randomly) as reference for current study, relevant for this outcome measure. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 44 | 44
Percentage of participants
  PMB80 (A22): number analyzed (Participants) | 44 | 43
  PMB80 (A22) | 75.0 [59.7 to 86.8] | 95.3 [84.2 to 99.4]
  PMB2001 (A56) | 90.9 [78.3 to 97.5] | 100.0 [92.0 to 100.0]
  PMB2948 (B24) | 70.5 [54.8 to 83.2] | 81.8 [67.3 to 91.8]
  PMB2707 (B44): number analyzed (Participants) | 43 | 42
  PMB2707 (B44) | 79.1 [64.0 to 90.0] | 92.9 [80.5 to 98.5]

3. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions (redness, swelling, and pain) at the site of investigational product administration were recorded in electronic diary (e-diary). Redness and swelling were measured and recorded in caliper units. Each caliper unit = 0.5 centimeter (cm). Redness and swelling were graded as mild (more than [>]2.0 to 5.0cm), moderate (>5.0 to 10.0cm) and severe (>10.0cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity).
Time Frame: Within 7 Days after Vaccination 1 (Vaccination 1 on Day 1/Month 0)
Population: B1971060: Vaccination 1 safety set included all participants who received the first dose of study intervention at Visit 1 and for whom safety information was available from Visit 1 to prior to Visit 3. B1971057: Historical data of the age- and sex-matched healthy participants (selected randomly) as reference for current study, relevant for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants
  Redness: Any | 18.9 [9.4 to 32.0] | 11.8 [4.4 to 23.9]
  Redness: Mild | 5.7 [1.2 to 15.7] | 5.9 [1.2 to 16.2]
  Redness: Moderate | 9.4 [3.1 to 20.7] | 3.9 [0.5 to 13.5]
  Redness: Severe | 3.8 [0.5 to 13.0] | 2.0 [0.0 to 10.4]
  Swelling: Any | 22.6 [12.3 to 36.2] | 11.8 [4.4 to 23.9]
  Swelling: Mild | 7.5 [2.1 to 18.2] | 7.8 [2.2 to 18.9]
  Swelling: Moderate | 15.1 [6.7 to 27.6] | 3.9 [0.5 to 13.5]
  Swelling: Severe | 0 [0.0 to 6.7] | 0 [0.0 to 7.0]
  Pain at injection site: Any | 86.8 [74.7 to 94.5] | 80.4 [66.9 to 90.2]
  Pain at injection site: Mild | 41.5 [28.1 to 55.9] | 47.1 [32.9 to 61.5]
  Pain at injection site: Moderate | 32.1 [19.9 to 46.3] | 33.3 [20.8 to 47.9]
  Pain at injection site: Severe | 13.2 [5.5 to 25.3] | 0 [0.0 to 7.0]

4. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions (redness, swelling, and pain) at the site of investigational product administration were recorded in electronic diary (e-diary). Redness and swelling were measured and recorded in caliper units. Each caliper unit = 0.5 cm. Redness and swelling were graded as mild (>2.0 to 5.0cm), moderate (>5.0 to 10.0cm) and severe (>10.0cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity).
Time Frame: Within 7 Days after Vaccination 2 (Vaccination 2 at Month 6)
Population: B1971060: Vaccination 2 safety set included all participants who received the second dose of study intervention at Visit 3 and for whom safety information was available from Visit 3 up to and including Visit 4. B1971057: Historical data of the age- and sex-matched healthy participants (selected randomly) as reference for current study, relevant for this outcome measure. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 45 | 43
Percentage of participants
  Redness: Any | 20.0 [9.6 to 34.6] | 7.0 [1.5 to 19.1]
  Redness: Mild | 6.7 [1.4 to 18.3] | 2.3 [0.1 to 12.3]
  Redness: Moderate | 11.1 [3.7 to 24.1] | 4.7 [0.6 to 15.8]
  Redness: Severe | 2.2 [0.1 to 11.8] | 0 [0.0 to 8.2]
  Swelling: Any | 26.7 [14.6 to 41.9] | 4.7 [0.6 to 15.8]
  Swelling: Mild | 13.3 [5.1 to 26.8] | 0 [0.0 to 8.2]
  Swelling: Moderate | 13.3 [5.1 to 26.8] | 4.7 [0.6 to 15.8]
  Swelling: Severe | 0 [0.0 to 7.9] | 0 [0.0 to 8.2]
  Pain at injection site: Any | 93.3 [81.7 to 98.6] | 60.5 [44.4 to 75.0]
  Pain at injection site: Mild | 44.4 [29.6 to 60.0] | 30.2 [17.2 to 46.1]
  Pain at injection site: Moderate | 35.6 [21.9 to 51.2] | 27.9 [15.3 to 43.7]
  Pain at injection site: Severe | 13.3 [5.1 to 26.8] | 2.3 [0.1 to 12.3]

5. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days After Vaccination 1
Description: Systemic events included: fever, fatigue, headache, chills, muscle pain, joint pain, vomiting, and diarrhea. Fever classified as =>38.0 degree Celsius (C), 38.0-38.4, >38.4-38.9, >38.9 40.0 and >40.0-degree C. Fatigue, headache, chills, muscle pain and joint pain graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily activity). Vomiting graded as mild (1-2 times in 24 hours [hrs]), moderate (>2 times in 24 hrs) and severe (required intravenous [IV] hydration). Diarrhea graded as mild (2-3 loose stools in 24 hrs), moderate (4-5 loose stools in 24 hrs) and severe (=>6 in 24 hrs).
Time Frame: Within 7 Days after Vaccination 1 (Vaccination 1 on Day 1/Month 0)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants
  Fever: =>38.0 degree C | 3.8 [0.5 to 13.0] | 2.0 [0.0 to 10.4]
  Fever: 38.0 to 38.4 degree C | 1.9 [0.0 to 10.1] | 0 [0.0 to 7.0]
  Fever: >38.4 to 38.9 degree C | 0 [0.0 to 6.7] | 2.0 [0.0 to 10.4]
  Fever: >38.9 to 40.0 degree C | 1.9 [0.0 to 10.1] | 0 [0.0 to 7.0]
  Fever: >40.0 degree C | 0 [0.0 to 6.7] | 0 [0.0 to 7.0]
  Fatigue: Any | 54.7 [40.4 to 68.4] | 51.0 [36.6 to 65.2]
  Fatigue: Mild | 26.4 [15.3 to 40.3] | 39.2 [25.8 to 53.9]
  Fatigue: Moderate | 22.6 [12.3 to 36.2] | 11.8 [4.4 to 23.9]
  Fatigue: Severe | 5.7 [1.2 to 15.7] | 0 [0.0 to 7.0]
  Headache: Any | 41.5 [28.1 to 55.9] | 29.4 [17.5 to 43.8]
  Headache: Mild | 18.9 [9.4 to 32.0] | 25.5 [14.3 to 39.6]
  Headache: Moderate | 18.9 [9.4 to 32.0] | 2.0 [0.0 to 10.4]
  Headache: Severe | 3.8 [0.5 to 13.0] | 2.0 [0.0 to 10.4]
  Chills: Any | 15.1 [6.7 to 27.6] | 19.6 [9.8 to 33.1]
  Chills: Mild | 11.3 [4.3 to 23.0] | 17.6 [8.4 to 30.9]
  Chills: Moderate | 1.9 [0.0 to 10.1] | 2.0 [0.0 to 10.4]
  Chills: Severe | 1.9 [0.0 to 10.1] | 0 [0.0 to 7.0]
  Muscle Pain: Any | 26.4 [15.3 to 40.3] | 23.5 [12.8 to 37.5]
  Muscle Pain: Mild | 15.1 [6.7 to 27.6] | 11.8 [4.4 to 23.9]
  Muscle Pain: Moderate | 9.4 [3.1 to 20.7] | 9.8 [3.3 to 21.4]
  Muscle Pain: Severe | 1.9 [0.0 to 10.1] | 2.0 [0.0 to 10.4]
  Joint Pain: Any | 22.6 [12.3 to 36.2] | 19.6 [9.8 to 33.1]
  Joint Pain: Mild | 9.4 [3.1 to 20.7] | 11.8 [4.4 to 23.9]
  Joint Pain: Moderate | 9.4 [3.1 to 20.7] | 5.9 [1.2 to 16.2]
  Joint Pain: Severe | 3.8 [0.5 to 13.0] | 2.0 [0.0 to 10.4]
  Vomiting: Any | 1.9 [0.0 to 10.1] | 2.0 [0.0 to 10.4]
  Vomiting: Mild | 1.9 [0.0 to 10.1] | 2.0 [0.0 to 10.4]
  Vomiting: Moderate | 0 [0.0 to 6.7] | 0 [0.0 to 7.0]
  Vomiting: Severe | 0 [0.0 to 6.7] | 0 [0.0 to 7.0]
  Diarrhea: Any | 9.4 [3.1 to 20.7] | 11.8 [4.4 to 23.9]
  Diarrhea: Mild | 9.4 [3.1 to 20.7] | 5.9 [1.2 to 16.2]
  Diarrhea: Moderate | 0 [0.0 to 6.7] | 5.9 [1.2 to 16.2]
  Diarrhea: Severe | 0 [0.0 to 6.7] | 0 [0.0 to 7.0]

6. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days After Vaccination 2
Description: Systemic events included: fever, fatigue, headache, chills, muscle pain, joint pain, vomiting, and diarrhea. Fever classified as =>38.0 degree C, 38.0-38.4, >38.4-38.9, >38.9 40.0 and >40.0-degree C. Fatigue, headache, chills, muscle pain and joint pain graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily activity). Vomiting graded as mild (1-2 times in 24 hrs), moderate (>2 times in 24 hrs) and severe (required IV hydration). Diarrhea graded as mild (2-3 loose stools in 24 hrs), moderate (4-5 loose stools in 24 hrs) and severe (=>6 in 24 hrs).
Time Frame: Within 7 Days after Vaccination 2 (Vaccination 2 at Month 6)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 45 | 43
Percentage of participants
  Fever: =>38.0 degree C | 2.2 [0.1 to 11.8] | 2.3 [0.1 to 12.3]
  Fever: 38.0 to 38.4 degree C | 2.2 [0.1 to 11.8] | 0 [0.0 to 8.2]
  Fever: >38.4 to 38.9 degree C | 0 [0.0 to 7.9] | 2.3 [0.1 to 12.3]
  Fever: >38.9 to 40.0 degree C | 0 [0.0 to 7.9] | 0 [0.0 to 8.2]
  Fever: >40.0 degree C | 0 [0.0 to 7.9] | 0 [0.0 to 8.2]
  Fatigue: Any | 53.3 [37.9 to 68.3] | 41.9 [27.0 to 57.9]
  Fatigue: Mild | 24.4 [12.9 to 39.5] | 23.3 [11.8 to 38.6]
  Fatigue: Moderate | 24.4 [12.9 to 39.5] | 14.0 [5.3 to 27.9]
  Fatigue: Severe | 4.4 [0.5 to 15.1] | 4.7 [0.6 to 15.8]
  Headache: Any | 35.6 [21.9 to 51.2] | 30.2 [17.2 to 46.1]
  Headache: Mild | 6.7 [1.4 to 18.3] | 23.3 [11.8 to 38.6]
  Headache: Moderate | 22.2 [11.2 to 37.1] | 7.0 [1.5 to 19.1]
  Headache: Severe | 6.7 [1.4 to 18.3] | 0 [0.0 to 8.2]
  Chills: Any | 8.9 [2.5 to 21.2] | 14.0 [5.3 to 27.9]
  Chills: Mild | 4.4 [0.5 to 15.1] | 11.6 [3.9 to 25.1]
  Chills: Moderate | 2.2 [0.1 to 11.8] | 2.3 [0.1 to 12.3]
  Chills: Severe | 2.2 [0.1 to 11.8] | 0 [0.0 to 8.2]
  Muscle Pain: Any | 13.3 [5.1 to 26.8] | 11.6 [3.9 to 25.1]
  Muscle Pain: Mild | 4.4 [0.5 to 15.1] | 7.0 [1.5 to 19.1]
  Muscle Pain: Moderate | 8.9 [2.5 to 21.2] | 2.3 [0.1 to 12.3]
  Muscle Pain: Severe | 0 [0.0 to 7.9] | 2.3 [0.1 to 12.3]
  Joint Pain: Any | 20.0 [9.6 to 34.6] | 16.3 [6.8 to 30.7]
  Joint Pain: Mild | 6.7 [1.4 to 18.3] | 14.0 [5.3 to 27.9]
  Joint Pain: Moderate | 11.1 [3.7 to 24.1] | 0 [0.0 to 8.2]
  Joint Pain: Severe | 2.2 [0.1 to 11.8] | 2.3 [0.1 to 12.3]
  Vomiting: Any | 2.2 [0.1 to 11.8] | 0 [0.0 to 8.2]
  Vomiting: Mild | 2.2 [0.1 to 11.8] | 0 [0.0 to 8.2]
  Vomiting: Moderate | 0 [0.0 to 7.9] | 0 [0.0 to 8.2]
  Vomiting: Severe | 0 [0.0 to 7.9] | 0 [0.0 to 8.2]
  Diarrhea: Any | 8.9 [2.5 to 21.2] | 4.7 [0.6 to 15.8]
  Diarrhea: Mild | 6.7 [1.4 to 18.3] | 4.7 [0.6 to 15.8]
  Diarrhea: Moderate | 2.2 [0.1 to 11.8] | 0 [0.0 to 8.2]
  Diarrhea: Severe | 0 [0.0 to 7.9] | 0 [0.0 to 8.2]

7. Primary Outcome: Percentage of Participants Reporting Use of Antipyretic Medication Within 7 Days After Vaccination 1
Time Frame: Within 7 Days after Vaccination 1 (Vaccination 1 on Day 1/Month 0)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 34.0 [21.5 to 48.3] | 9.8 [3.3 to 21.4]

8. Primary Outcome: Percentage of Participants Reporting Use of Antipyretic Medication Within 7 Days After Vaccination 2
Time Frame: Within 7 Days after Vaccination 2 (Vaccination 2 at Month 6)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 45 | 43
Percentage of participants | 28.9 [16.4 to 44.3] | 7.0 [1.5 to 19.1]

9. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) During 30 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs excluded local reactions and systematic events.
Time Frame: 30 Days after Vaccination 1 (Vaccination 1 on Day 1/Month 0)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 26.4 [15.3 to 40.3] | 9.8 [3.3 to 21.4]

10. Primary Outcome: Percentage of Participants Reporting AEs During 30 Days After Vaccination 2
Description: as for outcome 9
Time Frame: 30 Days after Vaccination 2 (Vaccination 2 at Month 6)
Population: B1971060: Vaccination 2 safety set included all participants who received the second dose of study intervention at Visit 3 and for whom safety information was available from Visit 3 up to and including Visit 4. B1971057: Historical data of the age- and sex-matched healthy participants (selected randomly) as reference for current study, relevant for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 47 | 47
Percentage of participants | 12.8 [4.8 to 25.7] | 12.8 [4.8 to 25.7]

11. Primary Outcome: Percentage of Participants Reporting AEs During 30 Days After Any Vaccination
Description: as for outcome 9
Time Frame: 30 Days after any Vaccination
Population: B1971060: Safety set included all enrolled participants who received at least 1 dose of the study intervention and have safety data reported after vaccination. B1971057: Historical data of the age- and sex-matched healthy participants (selected randomly) as reference for current study, relevant for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 34.0 [21.5 to 48.3] | 17.6 [8.4 to 30.9]

12. Primary Outcome: Percentage of Participants Reporting AEs During the Vaccination Phase
Description: as for outcome 9
Time Frame: Vaccination Phase: From Vaccination 1 through one Month after Vaccination 2 (approximately 7 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 60.4 [46.0 to 73.5] | 41.2 [27.6 to 55.8]

13. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs) During 30 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect or that was considered to be an important medical event.
Time Frame: 30 Days after Vaccination 1 (Vaccination 1 on Day 1/Month 0)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 9.4 [3.1 to 20.7] | 0 [0.0 to 7.0]

14. Primary Outcome: Percentage of Participants Reporting SAEs During 30 Days After Vaccination 2
Description: as for outcome 13
Time Frame: 30 Days after Vaccination 2 (Vaccination 2 at Month 6)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 47 | 47
Percentage of participants | 0 [0.0 to 7.5] | 0 [0.0 to 7.5]

15. Primary Outcome: Percentage of Participants Reporting SAEs During 30 Days After Any Vaccination
Description: as for outcome 13
Time Frame: 30 Days after any Vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 9.4 [3.1 to 20.7] | 0 [0.0 to 7.0]

16. Primary Outcome: Percentage of Participants Reporting SAEs During the Vaccination Phase
Description: as for outcome 13
Time Frame: Vaccination Phase: From Vaccination 1 through 1 Month after Vaccination 2 (approximately 7 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 17.0 [8.1 to 29.8] | 0 [0.0 to 7.0]

17. Primary Outcome: Percentage of Participants Reporting SAEs During the Follow-up Phase
Description: as for outcome 13
Time Frame: Follow-up Phase: From 1 Month after Vaccination 2 through 6 Months after Vaccination 2 (approximately 5 Months)
Population: B1971060: Follow-up safety set included all participants who received at least 1 dose of study intervention and for whom safety information was available from after Visit 4 up to and including Visit 5. B1971057: Historical data of the age- and sex-matched healthy participants (selected randomly) as reference for current study, relevant for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 44 | 48
Percentage of participants | 4.5 [0.6 to 15.5] | 2.1 [0.1 to 11.1]

18. Primary Outcome: Percentage of Participants Reporting SAEs During the Entire Study
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect. Or that was considered to be an important medical event.
Time Frame: Entire Study: From Vaccination 1 through 6 Months after Vaccination 2 (approximately 12 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 18.9 [9.4 to 32.0] | 2.0 [0.0 to 10.4]

19. Primary Outcome: Percentage of Participants Reporting Medically Attended Adverse Event (MAEs) During 30 Days After Vaccination 1
Description: MAEs was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: 30 Days after Vaccination 1 (Vaccination 1 on Day 1/Month 0)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 20.8 [10.8 to 34.1] | 5.9 [1.2 to 16.2]

20. Primary Outcome: Percentage of Participants Reporting MAEs During 30 Days After Vaccination 2
Description: MAEs was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: 30 Days after Vaccination 2 (Vaccination 2 at Month 6)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 47 | 47
Percentage of participants | 12.8 [4.8 to 25.7] | 4.3 [0.5 to 14.5]

21. Primary Outcome: Percentage of Participants Reporting MAEs During 30 Days After Any Vaccination
Description: MAEs was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: 30 Days after any Vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 30.2 [18.3 to 44.3] | 9.8 [3.3 to 21.4]

22. Primary Outcome: Percentage of Participants Reporting MAEs During the Vaccination Phase
Description: MAEs was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Vaccination Phase: From Vaccination 1 through 1 Month after Vaccination 2 (approximately 7 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 54.7 [40.4 to 68.4] | 29.4 [17.5 to 43.8]

23. Primary Outcome: Percentage of Participants Reporting MAEs During the Follow-up Phase
Description: MAEs was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Follow-up Phase: From 1 Month after Vaccination 2 through 6 Months after Vaccination 2 (approximately 5 Months)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 44 | 48
Percentage of participants | 15.9 [6.6 to 30.1] | 10.4 [3.5 to 22.7]

24. Primary Outcome: Percentage of Participants Reporting MAEs During the Entire Study
Description: MAEs was defined as a nonserious AE that resulted in an evaluation at a medical facility.
Time Frame: Entire Study: From Vaccination 1 through 6 Months after Vaccination 2 (approximately 12 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 60.4 [46.0 to 73.5] | 31.4 [19.1 to 45.9]

25. Primary Outcome: Percentage of Participants Reporting Immediate AEs After Vaccination 1
Description: Immediate AE was defined as AE occurring within the first 30 minutes after study intervention administration.
Time Frame: 30 Minutes post Vaccination 1 (Vaccination 1 on Day 1/Month 0)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 0 [0.0 to 6.7] | 2.0 [0.0 to 10.4]

26. Primary Outcome: Percentage of Participants Reporting Immediate AEs After Vaccination 2
Description: Immediate AE was defined as AE occurring within the first 30 minutes after study intervention administration.
Time Frame: 30 Minutes post Vaccination 2 (Vaccination 2 at Month 6)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 47 | 47
Percentage of participants | 0 [0.0 to 7.5] | 0 [0.0 to 7.5]

27. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Condition (NDCMC) During the Vaccination Phase
Description: A NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: Vaccination Phase: From Vaccination 1 through 1 Month after Vaccination 2 (approximately 7 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 1.9 [0.0 to 10.1] | 0 [0.0 to 7.0]

28. Primary Outcome: Percentage of Participants With NDCMC During the Follow-up Phase
Description: as for outcome 27
Time Frame: Follow-up Phase: From 1 Month after Vaccination 2 through 6 Months after Vaccination 2 (approximately 5 Months)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 44 | 48
Percentage of participants | 0 [0.0 to 8.0] | 0 [0.0 to 7.4]

29. Primary Outcome: Percentage of Participants With NDCMC During the Entire Study
Description: as for outcome 27
Time Frame: Entire Study: From Vaccination 1 through 6 Months after Vaccination 2 (approximately 12 Months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 53 | 51
Percentage of participants | 1.9 [0.0 to 10.1] | 0 [0.0 to 7.0]

30. Primary Outcome: Mean Number of Days Participants Missed School or Work Because of AEs During the Vaccination Phase
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Vaccination Phase: From Vaccination 1 through 1 Month after Vaccination 2 (approximately 7 Months)
Population: B1971060: Safety set included all enrolled participants who received at least 1 dose of the study intervention and have safety data reported after vaccination. B1971057: Historical data of the age- and sex-matched healthy participants (selected randomly) as reference for current study, relevant for this outcome measure. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
Number analyzed (Participants) | 32 | 21
Days | 12.7 (7.6) | 2.5 (2.3)

ADVERSE EVENTS:
Time Frame: Local reactions, systemic events within 7 days of each vaccination; SAEs and Non-SAEs: From Day 1 of vaccination up to 6 months after last study vaccination (approximately 12 months)
Description: Same event may appear as both AE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. For study B1971057 MedDRA version 25.1 was used and for study B1971060 MedDRA version 26.0 was used.
Arm/Group | Trumenba (B1971060) | Trumenba (B1971057, Historical Age- and Sex-Matched Control)
All-Cause Mortality (participants affected / at risk) | 1/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 10/53 | 1/51
Other Adverse Events (participants affected / at risk) | 51/53 | 49/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trumenba (B1971060) (N=53) | Trumenba (B1971057, Historical Age- and Sex-Matched Control) (N=51)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 4 (8) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trumenba (B1971060) (N=53) | Trumenba (B1971057, Historical Age- and Sex-Matched Control) (N=51)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3)
Headache (HEADACHE) (Nervous system disorders) | 25 (38) | 21 (28)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Periorbital swelling (Eye disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 8 (9) | 7 (8)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (VOMITING) (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 14 (19) | 6 (9)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 14 (21) | 13 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 16 (20) | 14 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 5 (5) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otitis media bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Tonsillitis (Infections and infestations) | 4 (4) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (5)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Urethritis mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Secondary hypertension (Vascular disorders) | 1 (1) | 0 (0)
Chills (CHILLS) (General disorders) | 11 (12) | 11 (16)
Fatigue (General disorders) | 1 (1) | 2 (2)
Fatigue (FATIGUE) (General disorders) | 31 (53) | 27 (44)
Injection site pain (General disorders) | 0 (0) | 2 (2)
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 48 (88) | 45 (67)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (FEVER) (General disorders) | 2 (3) | 2 (2)
Swelling (SWELLING) (General disorders) | 17 (24) | 7 (8)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT04893811/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT04893811/SAP_001.pdf